CLINICAL TRIAL: NCT07191171
Title: Impact of Dysbiosis-inducing Drugs on Effectivity of Immune Checkpoint Inhibitor in Non-small Cell Lung Cancer Patients: a Retrospective Study
Brief Title: Impact of Dysbiosis-inducing Drugs on Effectivity of Immune Checkpoint Inhibitor in Non-small Cell Lung Cancer Patients
Acronym: ICI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9540
Record Dates: First submitted 2025-04-07; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-04

CONDITIONS: Dysbiosis
Keywords: Dysbiosis; Lung cancer; Non-small cell lung cancer; Intestinal microbiota; Immunotherapy
MeSH Terms: conditions — Dysbiosis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cancer in France in terms of mortality. The prognosis of the disease is closely correlated with the diagnostic stage and the majority of patients are diagnosed at a metastatic stage. The arrival of immunotherapy has made it possible to change the therapeutic paradigm by significantly improving the survival of metastatic patients. Despite this progress, only 20 to 30% of patients respond to immunotherapy. The search for predictive factors of response to or resistance to these drugs is of major importance for better patient selection. Among these factors, the intestinal microbiota appears to be closely correlated with the response to immunotherapy via the education of adaptive anticancer immunity. Thus, several bacterial species have been associated with patient survival or disease progression. Interestingly, the abundance of these same bacteria can be modulated by certain drugs co-prescribed with immunotherapy. These dysbiotic treatments or those leading to a significant modification of the composition of the intestinal microbiota could then modulate the response to immunotherapy and therefore patient survival. The objective of this study is therefore to objectify the impact of several therapeutic classes modifying the intestinal microbiota initiated in the 90 days preceding D1 of immunotherapy on the survival of patients with locally advanced (stage III-C) or metastatic (stage IV) non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Confirmed diagnosis of NSCLC
* Stage IV or stage III-C NSCLC
* Immunotherapy treatment

Exclusion Criteria:

* Refusal to reuse data for scientific research purposes
* Minor patient
* Disease stage below stage III-C
* Patient included in a clinical trial with an unknown randomization arm (double-blind study)
* Lack of relevant data on concomitant treatments, biology, or clinical outcomes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) with confirmed diagnosis of NSCLC stage IV or stage III-C NSCLC and under imunotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 90 days preceding D1 of immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - CHU de Strasbourg - France, Strasbourg, France